CLINICAL TRIAL: NCT06314594
Title: The Individualized Stepwise Treatment Mode of Adolescent Idiopathic Scoliosis Based on Transformer Learning Algorithm
Brief Title: The Individualized Stepwise Treatment Mode of Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024KY920
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-03

CONDITIONS: Adolescent Scoliosis
MeSH Terms: interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): Conventional treatment
- intervention (Experimental): Using paradigms based on transfer learning and semi-supervised learning, using multiple learning methods, transformer image classification algorithms and other mathematical methods, an early warning model and stepped treatment model for adolescent scoliosis were developed and verified, and a cost-effectiveness analysis was conducted at the same time.
  Interventions: Procedure: Conventional treatment; Behavioral: intervention treatment

INTERVENTIONS:
Procedure: Conventional treatment — Patients will randomly assigned to routine treatment group (control group) and individualized treatment model group (intervention group). All patients will observed and intervened for 4 months. Patients in the control treatment group will follow the treatment plan in the 2016SOSORT guidelines
  Arms: intervention
Behavioral: intervention treatment — Patients will be input into the health management platform. The optimal treatment scheme will be then determined through data calculation and sent to individuals (or their families) or schools for implementation under the guidance of the platform. It is important to note that the specific treatment plan varied from person to person. Patients were observed and intervened for a period of 4 months.
  1. Massage therapy
  2. Posture guidance
  3. Schroeder's gymnastics therapy
  4. Bioelectric stimulation therapy
  Arms: intervention

SUMMARY:
Based on the risk factors affecting adolescent scoliosis found in the previous social survey, this project adopts the paradigm based on transfer learning and semi-supervised learning, and uses mathematical methods such as multiple learning methods and Transformer image classification algorithms to develop and verify the early warning model and stepped treatment model of adolescent scoliosis, and conducts cost-effect analysis.

DETAILED DESCRIPTION:
This study intends to build a standard system for the prevention and treatment of scoliosis in adolescents, do a good job in school health education and prevention and control work in school, comprehensively strengthen the construction of the prevention and control system of spondylosis, improve the ability of professionals in medical institutions, and give full play to the role of home-school-medical in the prevention and control of abnormal spinal curvature in children Firstly, relying on the investigation report, we independently develop the software platform and physical device for measuring, preventing and correcting scoliosis. Secondly, we use a series of prevention and control advantages to change from passive to active. Based on the Internet and big data technology, we integrate Western medicine data management and monitoring technology to establish the characteristics of the disease General disease information (personal history, family history, solar terms, climate and environment detection indicators, etc.) as one of the health management platform, the management platform set up health archives disease risk early warning health intervention and health promotion education follow-up management system management data quality control review data analysis and visualization 9 modules, respectively set up a management platform patient-side physician side and management background 3 parts through sampling investigation clinical research, break the medical school barriers, to build a personalized step treatment model for adolescent scoliosis.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of moderate and mild AIS, with a Cobb angle measuring less than 45°;
2. The age range of 12 to 16 years old;
3. Participants are required to have no history of mental illness, possess normal communication skills, and be proficient in reading and writing;
4. Signed informed consent by the patient or their family.

Exclusion Criteria:

Patients who fulfill any of the following conditions will be excluded a clear history of inducement, such as diseases caused by trauma, surgery, cognitive impairment, severe dysfunction of heart, liver, kidney and other organs, and malignant tumors, immune diseases and other malignant diseases.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Cobb angles | 4 months before the intervention and 4 months after the intervention
  X-rays were used to check the number of Cobb angles before and 4 months after the intervention to observe the improvement of scoliosis
Accuracy of new screening modalities | 4 months before and after the intervention, 4 months after the end of the intervention, and 8 months after the end of the intervention
  The new screening method "general examination + forward flexion test + scoliosis measuring instrument" was used for examination, and the data results before and 4 months after intervention were compared with the X-ray examination results to verify its accuracy.
Hamilton Depression Volume | 4 months before and after the intervention, 4 months after the end of the intervention, and 8 months after the end of the intervention
  Depression status was rated using the Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Xinyun Dr Li, doctor, Principal Investigator — hangzhou medical colleage
Locations (1):
- the Affiliated Zhejiang Provincial People's Hospital to Hangzhou Medical College., Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No